CLINICAL TRIAL: NCT03289429
Title: Comparative Study of the Antiarrhythmic and Cardioprotective Effects of Atorvastatin Versus Magnesium Sulfate in Cardiac Valve Replacement Surgery
Brief Title: Antiarrhythmic and Cardioprotective Effects of Atorvastatin Versus Magnesium Sulfate in Cardiac Valve Replacement Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, FATMA NABIL AHMED MOHAMED, Assistant lecturer of anesthesia and intensive care, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Statin and Magnesium
Record Dates: First submitted 2017-09-15; First posted 2017-09-21 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Arrhythmias
Keywords: Atorvastatin; Magnesium sulfate; POAF; Cardiac; Valve
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Atorvastatin; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Atorvastatin (Experimental): Atorvastatin and intravenous placebo
  Interventions: Drug: Atorvastatin; Other: intravenous placebo
- Magnesium sulfate (Experimental): Magnesium sulfate and tablets placebo
  Interventions: Drug: Magnesium Sulfate; Other: tablets placebo
- Control (Placebo Comparator): intravenous placebo and tablet placebo
  Interventions: Other: intravenous placebo; Other: tablets placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin in a dose of 80 mgs, twelve hours preoperatively, two hours preoperatively, and on the 2nd, 3rd, 4th and 5th postoperative days.
  Arms: Atorvastatin
Drug: Magnesium Sulfate — Magnesium sulfate: ( 3 grams dissolved in 100 mL of isotonic saline to be infused over 2 hours) twelve hours preoperatively, within the first hour of ICU arrival, and on the 2nd and 3rd postoperative days.
  Arms: Magnesium sulfate
Other: intravenous placebo — 100 mL of isotonic saline (to be infused over 2 hours) twelve hours preoperatively, within the first hour of ICU arrival, and on the 2nd and 3rd postoperative days.
  Arms: Atorvastatin; Control
Other: tablets placebo — Placebo tablets: twelve hours preoperatively, two hours preoperatively, and on the 2nd, 3rd, 4th and 5th postoperative days.
  Arms: Control; Magnesium sulfate

SUMMARY:
This study aims to compare the antiarrhythmic and cardioprotective effects of Atorvastatin versus Magnesium Sulfate after Cardiac valve Replacement Surgery

DETAILED DESCRIPTION:
Arrhythmia is a common complication after cardiac valve surgery. Postoperative atrial fibrillation (POAF) is the most common type of arrhythmia after cardiac surgery. It has different leading causes, including myocardial injury, inadequate myocardial protection, the effect of cardiopulmonary bypass, and electrolyte imbalance. Beta blockers, amiodarone, and magnesium sulfate are used for the management of POAF.

Statin is used commonly for its lipid lowering action, however, some studies shows that statin has powerful pleiotropic effects including its antiarrhythmic effect.

This study aims to compare the antiarrhythmic and cardioprotective effects of Atorvastatin versus magnesium sulfate after cardiac replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing isolated valvular replacement surgery.
* Preoperative rhythm: Sinus rhythm.
* Preoperative troponin I < 0.01 ng/mL.
* Normal lipid profile.
* White blood cells (4-11 X 103/mm3).
* Preoperative C-reactive protein < 3 mg/L.

Exclusion Criteria:

* History of atrial fibrillation.
* Any degree of heart block or patients with implanted pacemaker.
* Prior use of Antiarrhythmic drugs.
* Preoperative lipid lowering therapy (e.g statins) during the last 3 months.
* Previous treatment with any type of magnesium containing supplementation (the week before the intervention).
* Underlying heart failure or Left ventricular ejection fraction < 0.3.
* Previous myocardial infarction.
* Diabetes or other metabolic disorders.
* Renal diseases.
* Hepatic dysfunction.
* Underlying thyroid problems (hypo/hyperthyroidism).
* Underlying inflammatory disease (active or controlled)
* Immunosuppressive and anti-inflammatory medications for the treatment of coexisting conditions.
* Psychological disorders,
* Emergency cardiac surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2017-09-24 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative atrial fibrillation | Five days
  The occurrence of postoperative atrial fibrillation (POAF)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt